CLINICAL TRIAL: NCT06052683
Title: A Randomized Trial Evaluating Toxicity of Stereotactic Body Radiotherapy (SBRT) and Low-dose Rate Brachytherapy (LDRB) in Localized Prostate Cancer.
Brief Title: A Trial Evaluating Toxicity of SBRT and LDRB in Localized Prostate Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRT vs LDR-BT
Record Dates: First submitted 2023-09-08; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Low-dose rate brachytherapy (LDRB); Stereotactic Body RadioTherapy (SBRT)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: For the pilot study, patients will be randomized to receive one of the following treatments to a planned sample size of 48 patients. 24 patients will be randomized in each treatment arms. Once the pilot study will be completed, the investigators will conduct the large-scale research study enrolling 208 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Dose Rate Brachytherapy to the prostate using Iodine-125 seed implant (Active Comparator): Low-Dose Rate Brachytherapy to the prostate using Iodine-125 seed implant to a total dose of 144 Gy.
  Interventions: Radiation: Low-Dose Rate Brachytherapy to the prostate using Iodine-125 seed implant
- Stereotactic Body Radiation Therapy to the prostate (Experimental): Stereotactic Body Radiation Therapy to the prostate using 36.25 Gy in 5 fractions.
  Interventions: Radiation: Stereotactic Body Radiation Therapy to the prostate

INTERVENTIONS:
Radiation: Low-Dose Rate Brachytherapy to the prostate using Iodine-125 seed implant — Low-dose rate brachytherapy with Iodine-125 to a total dose of 144 Gy
  Arms: Low-Dose Rate Brachytherapy to the prostate using Iodine-125 seed implant
Radiation: Stereotactic Body Radiation Therapy to the prostate — Prostate Stereotactic Body Radiation Therapy using 36.25 Gy in 5 fractions
  Arms: Stereotactic Body Radiation Therapy to the prostate

SUMMARY:
The goal of this clinical trial is to compare SBRT (Stereotactic Body RadioTherapy) to LDRB (Low-Dose Rate Brachytherapy with Iodine-125 seed implant) in patients with low and favourable intermediate-risk prostate cancer. The two main questions it aims to answer are :

1. Does SBRT (Stereotactic Body RadioTherapy) for low and intermediate risk prostate cancer patients will result in less genito-urinary (GU) and gastro-intestinal (GI) toxicities than LDRB (Low-Dose Rate Brachytherapy)?
2. Does prostate cancer patients treated by SBRT have a better quality of life than patients treated by LDRB

No randomized trial has yet compared LDRB to SBRT head to head.

DETAILED DESCRIPTION:
Low-dose rate brachytherapy (LDRB) using Iodine-125 seed implant is known to be an effective definitive treatment for patients with low and favourable intermediate-risk prostate cancer. Mature data from Canadian institutions reported a biochemical progression-free survival as high as 90-95% at 5-10 years for patients with low and intermediate risk disease.

Prostate Stereotactic Body Radiotherapy (SBRT) as a single modality is a promising alternative to LDRB in low and favourable intermediate-risk prostate cancer. Some studies have shown the feasibility and efficacy of SBRT with low to intermediate risk-prostate cancer with 5-7 years PSA-progression-free survival really high (89,8% to 97,1% at a median follow-up of 5-7 years) [PSA: Prostate-Specific Antigen]. No randomized trial has yet compared LDRB to SBRT head to head.

Acute urinary toxicity is not trivial: a few studies have shown correlation between late urinary toxicity and the presence of acute urinary toxicity in patients treated with LDRB. Our research hypothesis is that SBRT for low and intermediate risk will result in fewer toxicities at the genito-urinary and the gastro-intestinal levels after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within the last 8 months. Patients on active surveillance with evidence of disease progression are eligible to the protocol as long as they meet the eligibility criteria and have a recent prostate biopsy (within 8 months).
* Low-risk and favourable intermediate-risk prostate cancer patients are eligible according to the following definitions:

Low-risk disease defined as: Clinical stage T1-T2a and Gleason 6 and PSA ≤ 10 ng/mL

Favourable intermediate-risk cancer defined by a single NCCN intermediate risk factor:

[NCCN : National Comprehensive Cancer Network]

1. Clinical stage T2b
2. PSA > 10 but ≤ 20 ng/mL
3. Gleason 7 (3+4)

Lymph node evaluation by either computed tomography (CT) or magnetic resonance imaging (MRI) is optional and is left at the discretion of the treating physician.

* Age ≥ 18 years
* Eastern Cooperative Oncology Group performance status 0-1
* Patient considered medically fit for LDR brachytherapy
* Prostate volume ≤ 60 cc, measured by Trans-Rectal UltraSound (TRUS), CT or MRI, within the last 6 months.
* International Prostate Symptom Score (IPSS) ≤ 20 (alpha blockers allowed)
* No alpha reductase inhibitors use within two weeks of randomization
* No hormonal therapy is accepted
* Patients must provide a study-specified informed consent form prior to study entry.
* Patients must be willing and able to complete the EPIC-26, IPSS and SHIM questionnaires.

[EPIC-26: Expanded Prostate Cancer Index Composite score ; SHIM: Sexual Health Inventory for Men questionnaire].

Exclusion Criteria:

* Clinical or radiological evidence of metastatic disease or nodal involvement.
* Clinical stage ≥ T2b.
* Gleason score ≥ 4 + 3.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 3 years.
* Prior radical surgery for carcinoma of the prostate, or prior TURP (Trans-Urethral Resection of the Prostate).
* Prior pelvic radiotherapy or prior radiotherapy that would result in overlap of radiation fields.
* Prior chemotherapy for prostate cancer, or prior chemotherapy within the last 3 years.
* Prior cryosurgery of the prostate.
* Prior or current bleeding diathesis making fiducial placement or brachytherapy procedure unsafe.
* Previous androgen deprivation therapy within 6 months of the registration.
* Bilateral hip prostheses
* Any severe active comorbidity, laboratory abnormality, psychiatric illnesses, active or uncontrolled infections, serious illnesses or medical conditions that would prevent the patient from participating or to be managed according to the protocol (according to investigator's decision). Such examples includes active inflammatory bowel disease, significant urinary symptoms,

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 208 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Evaluation according to the CTCAE version 4 to assess non-inferiority of SBRT compared to LDRB. | 1, 3, 6, 9, 12, 18, 24 months after end of treatment and yearly after, up to 5 years.
  Number of toxicities events assessed

SECONDARY OUTCOMES:
Quality of life issues in patients with prostate cancer | At baseline, 3, 6, 9, 12, 18 and 24 months and then yearly after, up to 5 years.
  Expanded Prostate Cancer Index Composite score (EPIC-26 questionnaire). In general terms, a higher score represents a better health-related quality of life.
Urinary function | At baseline, 1, 3, 6. 9, 12, 18, 24 and 36 months after the procedure
  International Prostate Symptom Score (IPSS score). The IPSS score is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Absolute PSA nadir to evaluate biochemical disease free survival. | PSA measurement every 3 months after the procedure, during the first 3 years and then every 6 months, up to 5 years
  PSA measurements

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Thibault, MD, FRCPC, Study Chair — CHU de Québec-Université Laval
Locations (1):
- Centre Intégré de Cancérologie, CHU de Québec-Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No